CLINICAL TRIAL: NCT01857895
Title: An Open-Label Exploratory Study to Investigate the Feasibility of Administering Exenatide by Continuous Subcutaneous Infusion to Healthy Subjects
Brief Title: Feasibility Study of Exenatide by Continuous Subcutaneous Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200016
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: Nausea; subcutaneous infusion; exenatide
MeSH Terms: conditions — Obesity; Nausea | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide infusion in Part A (Experimental): Subjects in Part A will receive exenatide as a subcutaneous infusion at a constant rate for 24 hours.
  Interventions: Drug: Exenatide
- Exenatide infusion in Part B (Experimental): Subjects in Part B will receive exenatide with daily increases in the infusion rate.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Prefilled pen containing 2.4 mL of drug will be transferred into MiniMed Paradigm Real-Time Revel device for subcutaneous infusion.

SUMMARY:
This is an open-label study to investigate the feasibility of administering exenatide by continuous subcutaneous infusion to healthy subjects. Study will consist of two parts i.e. Part A and B. In Part A 2 healthy subjects will receive exenatide infusion over 24 hours followed by a follow-up visit 10 to 14 days after discharge from clinic. In Part B approximately 6 healthy subjects will receive subcutaneous infusions of exenatide for maximum of 7 days followed by a follow-up visit 10 to 14 days after discharge from clinic.

ELIGIBILITY:
Inclusion Criteria

* Male/females aged between 18 and 60 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and objectives.
* Body Mass Index within the range 18 to 35 kilograms/meter squared (kg/m^2) inclusive.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone > 40 milli international unit/mililiter (mL) and estradiol <40 picogram/mL (<147 picomoles/Liter) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.
* Child-bearing potential females must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until follow up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Based on QT interval corrected for heart rate (QTc) of single electrocardiogram (ECG): QTc by Fridericia's formula <450 millisecond (msec).
* Aspartate aminotransferase and Alanine aminotransferase <2x upper limit of normal (ULN); alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria

* Subjects with a personal or family history of thyroid carcinoma or Type 2 Familial Endocrine Neoplasia.
* History of uncorrected thyroid dysfunction or an abnormal thyroid functions as assessed by thyroid stimulating hormones.
* Subjects with a history of severe gastrointestinal disease, or abnormal renal function.
* Subjects with previous exposure to a Glucagon-like peptide-1 mimetic.
* History of chronic or acute pancreatitis. Note: Subjects with a lipase value above 1.5X ULN at screening are excluded.
* Current or chronic history of liver disease, or hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy.

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* A subject with a positive urine cotinine test result will be excluded from the study unless in the judgment of the Investigator the subject will be able to abstain from using tobacco for the duration of the in-house period of the study.
* A positive test for human immuno virus antibody.

Other Criteria

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2013-11-01 (Actual)

PRIMARY OUTCOMES:
Characterization of interruptions or deviations from prescribed exenatide infusion in Part A | 2 days
  To investigate the feasibility of administering exenatide via continuous subcutaneous infusion
Characterization of interruptions or deviations from prescribed exenatide infusion in Part B | 8 days
  To investigate the feasibility of administering exenatide via continuous subcutaneous infusion
Infusion rate adjustments when nausea/vomiting occurs in Part B | 8 days
  To investigate the feasibility of administering exenatide via continuous subcutaneous infusion. Infusion rate adjustment will be done to achieve tolerable infusion rate when nausea/vomiting occurs
Number of participants with adverse events (AEs) in Part A | 17 days
  AEs will be collected from the Day -1 and until the follow-up contact. AE data will be collected to evaluate the ability to monitor and maintain acceptable safety
Number of participants with AEs in Part B | 23 days
  AEs will be collected from the Day -1 and until the follow-up contact. AE data will be collected to evaluate the ability to monitor and maintain acceptable safety
Laboratory parameter assessment in Part A | 17 days
  Laboratory parameters include: hematology, clinical chemistry, and urinalysis
Laboratory parameter assessment in Part B | 23 days
  Laboratory parameters include: hematology, clinical chemistry, and urinalysis
Vital sign assessment in Part A | 17 days
  Vital signs measurement include: systolic and diastolic blood pressure, and pulse rate
Vital sign assessment in Part B | 23 days
  Vital signs measurement include: systolic and diastolic blood pressure, and pulse rate

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of exenatide in Part A | PK samples will be collected at pre-dose, and at 0.5, 1, 2, 4, 6, 10, 14, 24, and 26 hours post dose.
  PK parameters include: area under concentration time curve from time 0 to 24 hours (AUC0 to24), maximum observed concentration from time 0 to 24 hours (Cmax0 to 24), and average concentration from time 0 to 24 hours (Cavg0 to 24) versus time
Pharmacokinetic (PK) profile of exenatide in Part B | 8 days
  PK parameters include: AUC0-24, Cmax0 to 24, and Cavg0 to 24 versus time for each of 7 days and AUC0 to 168, Cmax0 to 168, and Cavg0 to 168 versus time over entire infusion period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Vlasakakis G, Johnson SL, Lin J, Yao X, Gruenloh CJ, Chism JP, Nunez DJ. Pharmacokinetics and Tolerability of Exenatide Delivered by 7-Day Continuous Subcutaneous Infusion in Healthy Volunteers. Adv Ther. 2015 Jul;32(7):650-61. doi: 10.1007/s12325-015-0222-4. Epub 2015 Jul 10. PMID 26160357
- See also: Results for study 200016 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200016?search=study&study_ids=200016#rs
- Available data/document: Study Protocol: 200016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200016 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register